CLINICAL TRIAL: NCT06247514
Title: The Balanced and Empowered Eating (BEET) in Diabetes Feasibility Trial
Brief Title: The BEET Diabetes Feasibility Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-1891; K23DK134758 (NIH)
Record Dates: First submitted 2024-01-25; First posted 2024-02-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Disordered Eating Behaviors
Keywords: Type 2 diabetes; Disordered Eating Behaviors; Cognitive behavioral therapy; Diabetes distress; Depression; Anxiety; Diabetes self-efficacy
MeSH Terms: conditions — Disordered Eating Behavior; Diabetes Mellitus, Type 2; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility trial.
  BHPs will be randomized and trained to deliver the intervention or the comparator. They will be encouraged to deliver the programs as they typically would in a clinical setting while maintaining fidelity to session content.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The BEET Diabetes Program (Experimental): The BEET Diabetes program consists of 6 sessions that follow a sequence: the first 3-sessions weekly and the last 3-sessions every other week. These sessions help participants learn strategies and health behavior change through a self-monitoring form. Supporters (in this study, the BHPs) guide individuals through the program, maintain motivation, and facilitate appropriate goal-setting. The BEET Diabetes Program emphasizes treating disorder eating behaviors (DEBs) in the context of diabetes (i.e., psychoeducation on DEBs in diabetes, optimal daily glucose management, benefits of physical activity, and fruit and vegetable intake).
  Interventions: Behavioral: The BEET Diabetes Program
- Cognitive behavioral Therapy Guided Self-help (Active Comparator): The Cognitive Behavioral Therapy Guided Self-help consists of 6 sessions that follow a sequence: the first 3-sessions weekly and the last 3-sessions every other week. These sessions help participants learn strategies and health behavior change through a self-monitoring form. The CBTgsh program is delivered through the self-help book: "Overcoming Binge Eating" by Christopher G. Fairburn. Guided support sessions can be provided by personnel with no background training or knowledge of CBT or DEBs, as the book acts as the "expert."
  Interventions: Behavioral: Cognitive Behavioral Therapy Guided Self-Help

INTERVENTIONS:
Behavioral: The BEET Diabetes Program — The BEET Diabetes program is an adapted CBT program specifically designed to treat disordered eating and improve diabetes self-management. Participants receive support from BHPs to guide them through the program, maintain motivation, and facilitate appropriate goal setting.
  Other Names: The Balanced and Empowered Eating (BEET) In Diabetes Program
  Arms: The BEET Diabetes Program
Behavioral: Cognitive Behavioral Therapy Guided Self-Help — 6-session cognitive behavioral therapy delivered through the self-help book "Overcoming Binge Eating Self-help" by Christopher G. Fairburn.
  The manual focuses on reducing binge-eating episodes. Guided support sessions can be provided by personnel with no background training or knowledge of CBT or disordered eating behaviors, as the book acts as the "expert."
  Other Names: Overcoming Binge Eating by Christopher G. Fairburn
  Arms: Cognitive behavioral Therapy Guided Self-help

SUMMARY:
Disordered eating behaviors (DEBs, e.g., binge eating or restrictive eating) can significantly impact type 2 diabetes (T2D) self-management and engagement in treatment for diabetes. Managing DEBs is a treatment component in diabetes self-management; however, it is not often the primary focus, and trained behavioral health providers are inconsistently involved in comprehensive diabetes management. This study plans to pilot two behavior change programs for disordered eating in T2D and gather information on factors that predict successful adoption and implementation in real-world clinical settings.

DETAILED DESCRIPTION:
The study aims are:

Aim 1: The investigators will engage behavioral health providers (BHPs) to refine the Balanced and Empowered Eating in Diabetes (or the BEET Diabetes Program) for implementation in real-world settings. The rationale for engaging and collaborating with BHPs and practice stakeholders early in the research protocol is based on data that few evidence-based psychological programs have been successfully translated into clinical settings. Once the six BHPs are recruited, they will be randomized to receive training and deliver either the intervention (i.e., the BEET Diabetes Program) or the comparator, Cognitive Behavior Therapy (CBT). Then, the investigators will collaborate with the BHPs to refine the behavior change programs for implementation in their clinical settings.

Aim 2: The investigators will determine the reach and feasibility of the BEET Diabetes Program in real-world settings. After the intervention refinement period, BHPs will implement and deliver either the intervention or the comparator. To evaluate the adoption, implementation, and potential for maintenance of the BEET Diabetes Program in clinical settings, guided by the RE-AIM framework, the study staff will collect data from clinical leaders, providers and staff, and BHPs via REDCap surveys, observation of sessions delivered by BHPs (live or audio recorded sessions) following a detailed checklist, and data extraction on referral rates and provider adoption from the electronic medical record (e.g., gathering data on the number of referrals or orders submitted by providers in their clinic). The investigators will also conduct semi-structured, 60-minute interviews via Zoom to determine perceived program value and potential for maintenance and long-term use of the programs.

Aim 3: The investigators will estimate the effectiveness of the BEET Diabetes Program on patient-reported and clinical outcomes. This is a Phase IIb pilot study to examine research protocol feasibility, intervention acceptability, patient reach, and engagement and estimate intervention effectiveness to finalize the processes and procedures. Patients will be screened and recruited for the study by their BHP in this aim.

ELIGIBILITY:
Inclusion Criteria:

* T2DM diagnosis
* HbA1c ≥ 6.5
* Positive disordered eating screen: Scored ≥ 2 on the study pre-screen for Disordered Eating OR ≥2 on the Diabetes Eating Problems Survey-Revised (DEPS-R) question #2 (skipping meals), #8 (binge eating), or #15 (self-induced vomiting)

Exclusion Criteria:

* Pregnancy or planning to become pregnant in the next 12 months
* Limited cognitive capacity (e.g., dementia or developmental disorder)
* Less than a year of life expectancy
* Plans to leave the practice in the next year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Disordered Eating Behaviors (DEBs) - Change in Participant-Reported Outcomes (PROs) | At the end of the 6 CBT sessions (weekly or biweekly) and 4-weeks after program completion (time differs by practice, up to 6 months)
  Comparison of change in patient-reported outcomes around diabetes eating problems for participants with type 2 diabetes. The Diabetes Eating Problems Survey - Revised (DEPS-R) is a validated self-reported screening tool comprising 16 items that assess diabetes-specific eating issues. Participants will be asked about eating habits, diabetes control, insulin misuse, and other compensatory behaviors.
  Higher scores indicate greater eating disorder psychopathology. Scores greater than 20 indicate individuals with a level of disordered eating warranting further attention.

SECONDARY OUTCOMES:
Diabetes Distress - Change in Participant-Reported Outcome (PROs) | After completion of the 6 CBT sessions and 4-weeks after program completion (time differs by practice, up to 6 months)
  Comparison of change in patient-reported outcome around diabetes distress. Measured by the Diabetes Distress Scale-17 (DDS-17). The DDS-17 measures distress in four domains: emotional burden, interpersonal distress, physician-related distress, and regimen-related distress. The DDS is a 17-item self-report instrument. Each of the 17 items is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem." A score of < 2.0 was defined as little or no distress, 2.0-2.9 as moderate distress, and ≥ 3.0 as high distress.
Diabetes Self-Efficacy - Change in Participant-Reported Outcome (PROs) | After completion of the 6 CBT sessions and 4-weeks after program completion (time differs by practice, up to 6 months)
  The Diabetes Self-Efficacy Scale (DSES) is a brief assessment measuring confidence in self-management behaviors. DSES is a reliable and valid instrument for assessing self-efficacy related to diabetes self-management. The DSES has eight items answered on an eight-point Likert scale, ranging from 1 (not confident at all) to 10 (totally confident). The total DSES score ranges from 8 to 80, with higher scores indicating higher diabetes self-efficacy.
Depression - Change in Participant-Reported Outcome (PROs) | After completion of the 6 CBT sessions and 4-weeks after program completion (time differs by practice, up to 6 months)
  Comparison of change in patient-reported outcomes around depression measured by the Personal Health Questionnaire-8 (PHQ-8), an 8-item scale used for diagnostic and severity measures for depressive disorders in large clinical studies. PHQ-8 score ≥ 10 represents clinically significant depression.
Anxiety - Change in Participant-Reported Outcome (PROs) | After completion of the 6 CBT sessions and 4-weeks after program completion (time differs by practice, up to 6 months)
  Comparison of change in patient-reported outcomes around anxiety measured by the Generalized Anxiety Disorder Scale 7 (GAD-7), a widely used scale with 7 questions to assess symptoms of Generalized Anxiety Disorder. GAD-7 total score for the seven items ranges from 0 to 21, which are 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety.
Change in participant's HbA1c | Baseline, After completion of the 6 CBT sessions and 4-weeks after program completion (time differs by practice, up to 6 months)
  Comparison of change in participant's HbA1c levels in either intervention. Measured by Siemens DCA Vantage (Potassium Ferricyanide), it evaluates the average amount of glucose in the blood, measuring the percentage of glycated (glycosylated) hemoglobin. A decreased value indicates improvements in glucose functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Phoutdavone Phimphasone-Brady, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado